CLINICAL TRIAL: NCT05632861
Title: Efficacy and Safety of HuHuangLianzonggan Capsule in Subjects With Nonalcoholic steatoHEPAtitis: a Randomized, Double-blind, Placebo-controlled, Multi-center, Phase 2 tRial(HHL-HEPAR)
Brief Title: HuHuangLianzonggan Capsule in Subjects With Nonalcoholic Steatohepatitis: a Phase 2 tRial(HHL-HEPAR)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tasly Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TSL-TCM-HHLZGJN-NASH-Ⅱ
Record Dates: First submitted 2022-11-13; First posted 2022-12-01 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: NASH

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): HuHuangLianzonggan capsule, 4 pills, take orally after meals, 2 times a day
  Interventions: Drug: HuHuangLianzonggan capsule
- Placebo group (Placebo Comparator): HuHuangLianzonggan capsule placebo, 4 pills, take orally after meals, 2 times a day
  Interventions: Drug: HuHuangLianzonggan capsule placebo

INTERVENTIONS:
Drug: HuHuangLianzonggan capsule — HuHuangLianzonggan capsule, 4 pills(120 mg per pill), take orally after meals, 2 times a day for 12weeks
  Other Names: Experimental group
  Arms: Experimental group
Drug: HuHuangLianzonggan capsule placebo — HuHuangLianzonggan capsule placebo, 4 pills(120 mg per pill), take orally after meals, 2 times a day for 12weeks
  Other Names: Placebo group
  Arms: Placebo group

SUMMARY:
This study will evaluate the efficacy and safety and the best effective dose of HuHuangLianzonggan capsule in subjects with nonalcoholic steatohepatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 18-75 years of age inclusive(including boundary values).
2. Must have had a liver biopsy proven NASH within 6 months or in screening test. The following two requirements must be met at the same time: ① a non-alcoholic fatty liver disease (NAFLD) activity score (NAS) of ≥ 4 with at least a score of 1 in each of the following NAS components: Steatosis≥1, Lobular inflammation≥1, Ballooning degeneration≥1;② fibrosis stage 1 to 3.
3. Must have confirmation of ≥ 8% liver fat content on magnetic resonance imaging- proton density fat fraction (MRI-PDFF) at screening.
4. No alcohol consumption or history of excessive alcohol consumption: less than 210 g of ethanol per week for men and 140 g for women in the past 12 months.
5. Patients who are taking chronic drugs(including but not limited to antihypertensive drugs, antiatherogenic drugs, oral hypoglycemic drugs, insulin) need to have a steady dose for at least 3 months before liver biopsy.
6. Weight was stable(the change is no more than 5%) during the 6 months prior to Screening.
7. No attempt to change lifestyle (diet and/or exercise) during the 3 months prior to Screening.
8. Ability to understand the requirements of the study and willingness to provide written informed consent.
9. Have no pregnancy program and take effective contraceptive measures voluntarily.
10. Abide by the experimental protocol and cooperate with the data collection according to the researcher's judgment.

Exclusion Criteria:

1. Treatment with drugs that may cause non-alcoholic fatty liver disease (NAFLD) administered for at least 2 weeks within 12 months prior to qualifying liver biopsy (e.g. valproic acid, tamoxifen, methotrexate, amiodarone, oral corticosteroids, >5 mg/day of prednisone equivalent [one short (<2 weeks) course of oral corticosteroids, more than 3 months before the liver biopsy is allowed], or oestrogens [at doses greater than those used for contraception or hormone replacement]).
2. Documented causes of fatty liver disease other than NASH including, but not restricted to: HCV-associated fatty liver (genotype 3), hepatolenticular degeneration, autoimmune hepatitis, total parenteral nutrition, abetalipoproteinemia, lipoatrophy , Coeliac disease, Primary sclerosing cholangitis, Alpha-1-antitrypsin deficiency, Drug-induced liver disease.
3. Model for End-stage Liver Disease (MELD) score >12.
4. Histologically documented liver cirrhosis (fibrosis stage F4), history or current diagnosis of hepatocellular carcinoma HCC.
5. History of or planned liver transplant.
6. Viral hepatitis：Positive hepatitis A antibody，Positive hepatitis D antibody，Positive hepatitis E antibody，Positive hepatitis B surface antigen (HBsAg) ，Positive hepatitis C antibody.
7. Abnormal liver function as defined by Screening central laboratory evaluation of any of the following: ALT or AST >5 × ULN; Alkaline phosphatase (ALP) >2 × ULN; albumin below the lower limit of the normal range; total bilirubin level >1.5 × ULN (patients with a documented history of Gilbert's syndrome can be enrolled if the direct bilirubin is within normal reference range).
8. In patients who are not anticoagulated, INR ≥ 1.3 times ULN or other evidence of impaired coagulation.
9. Renal impairment measured as estimated Glomerular Filtration Rate (eGFR) value <30 mL/min/1.73 m2.
10. Patient currently receiving any approved treatment for NASH.
11. HbA1c ≥9% or fasting blood-glucose>13.9 mmol/L at Screening.
12. Diabetes mellitus other than type 2 (e.g. type 1, diabetes caused by drugs or chemicals, and immune-mediated diabetes).
13. Those who are underweight, of normal weight, or severely obese, i.e BMI<23 kg/m2 or BMI≥40 kg/m2.
14. Bariatric surgery or tumor surgery are not allowed within 5 years of the qualifying liver biopsy.
15. Uncontrolled hypertension (values ≥160/100 mm Hg) or hypotension（values <80/50 mmHg）.
16. Acute vascular events including ACS, stroke, peripheral vascular disease worsened, or any vascular/cardiac surgery within the 6 months prior to Screening.
17. Concomitant mental illness and poor condition control, which affects the signing of informed consent or presentation of adverse events.
18. Do not have a liver biopsy within the 6 months prior to Screening and refuse to take liver biopsy at Screening.
19. Allergic constitution, or allergic to the test drug or its ingredients.
20. Women who are pregnant or lactating.
21. Participate in clinical trials of other drugs within 3 months before screening.
22. The researchers did not consider it appropriate to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in hepatic fat fraction assessed by MRI-PDFF at week 12. | Week 12
Proportion of subjects with ≥ 30% relative fat reduction on MRI-PDFF at week 12. | Week 12

SECONDARY OUTCOMES:
Change from baseline in weight at week 4, 12. | Week 4, 12
Change from baseline in Body Mass Index (BMI) at week 4, 12. | Week 4, 12
Change from baseline in waist hip rate at week 4, 12. | Week 4, 12
Change from baseline in fasting blood glucose at week 4, 12. | Week 4, 12
Change from baseline in 2 hours postprandial hyperglycemia at week 4, 12. | Week 4, 12
Change from baseline in homeostasis model assessment-insulin resistance (HOMA-IR) at week 4, 12. | Week 4, 12
Change from baseline in Total Cholestrol (TC) at week 4, 12. | Week 4, 12
Change from baseline in triglyceride (TG) at week 4, 12. | Week 4, 12
Change from baseline in Low Density Lipoprotein Cholesterol (LDL-C) at week 4, 12. | Week 4, 12
Change from baseline in High Density Lipoprotein Cholesterol (HDL-C) at week 4, 12. | Week 4, 12
Change from baseline in Glycosylated hemoglobin A1c (HbA1c) at week 12. | Week 12
Change from baseline in Alanine aminotransferase (ALT) at week 4, 12. | Week 4, 12
Change from baseline in Aspartate aminotransferase (AST) at week 4, 12. | Week 4, 12
Change from baseline in total bilirubin (TBil) at week 4, 12. | Week 4, 12
Change from baseline in Cytokeratin18 (CK-18) at week 4, 12. | Week 4, 12
Change from baseline in N-terminal type Ⅲ collagen propeptide (Pro-C3) at week 4, 12. | Week 4, 12
Change from baseline in Fibrosis 4 score at week 4, 12. | Week 4, 12
Change from baseline in Chronic Liver Disease-NAFLD questionnaire (CLDQ-NAFLD) at week 4, 12. | Week 4, 12
Change from baseline in ferritin at week 4, 12. | Week 4, 12

CONTACTS AND LOCATIONS:
Locations (20):
- China (20):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The first affiliated hospital of Fujian medical university, Fuzhou, Fujian
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - The Third People's Hospital of Shenzhen, Shenzhen, Guangdong
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - The First People's Hospital of Lianyungang, Lianyungang, Jiangsu
  - The Affiliated Hospital of Nanjing University medical school，Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - The Second Hospital of Nanjing, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Tianjin Second People's Hospital, Tianjin, Tianjin Municipality
  - The Affiliated Hospital of Hangzhou Normal University, Hangzhou, Zhejiang
  - Ningbo Huamei Hospital, University of Chinese Academy of Sciences, Ningbo, Zhejiang
  - Ningbo Medical Center Lihuili Hospital, Ningbo, Zhejiang
  - Taizhou Municipal Hospital, Taizhou, Zhejiang
  - Rui'an People's Hospital, Wenzhou, Zhejiang